CLINICAL TRIAL: NCT06156384
Title: Prospective, Observational Study to Assess the Pain, Satisfaction, and Quality of Life of Patients Implanted With the FITBONE® Lengthening Nail
Brief Title: Study to Assess the Pain, Satisfaction, and Quality of Life of Patients With FITBONE® Lengthening Nail
Acronym: FitForFrance
Status: Recruiting | Type: Observational
Sponsor: Orthofix s.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: OCI_2301; 2023-A02702-43 (Other: ID-RCB number (France))
Record Dates: First submitted 2023-11-22; First posted 2023-12-05 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Leg Length Inequality
Keywords: Fitbone; LLD; Bone lengthening; Nail; Nailing; Intramedullary nailing; Intramedullary nail; Motorized Nail
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients aged ≥12 years with congenital or acquired lower limb discrepancy, greater than 30mm
  Interventions: Device: FITBONE® Lengthening Nail

INTERVENTIONS:
Device: FITBONE® Lengthening Nail — The patient is installed on a standard orthopaedic table, intramedullary reaming is performed through a metal working tube. The osteotomy is performed percutaneously and then an osteotome according to the postage-stamp technique. Once the FITBONE lengthening nail is placed in the desired location, it should be connected to the subcutaneous receiver. The receiver should be placed close enough to the skin surface to ensure the energy transfer from the external transmitter.
  After 5 to 10 days after surgery, the lengthening mechanism is operated by the patient, using the transmitter. An elongation of approximately 1 mm/day takes place. The attending physician determines the rhythm of lengthening in each case. When the desired elongation length is reached, the consolidation phase begins, which is necessary for bone regeneration. The FITBONE lengthening nail can be removed once the bone has consolidated, approximately one to one and a half years after implantation.

SUMMARY:
This study is a prospective observational non-interventional multi-centre cohort study of patients, 12 years or older, initiating a lower limb lengthening procedure with FITBONE and who have a length discrepancy of 30mm or more between the limbs.

The following parameters will be assessed for up to 24 months.

* Pain using the Visual Analog Scale (VAS), Patient Global Assessment (PGA) and Clinical Observer Global Assessment (COGA)
* Patient satisfaction using the Patient Global Impression of change (PGI-C) scale
* QoL using the 36-Item Short Form Survey/Paediatric Quality of Life Inventory (SF-36/PedsQL)

DETAILED DESCRIPTION:
The study period is 24 months post-surgery. Each patient's demographic data, medical history, any relevant concomitant medication, physical examination, range of motion data will be recorded using a standardized case record form after informed consent is provided and the healthcare provider completes a physical examination regarding the patient's conditions and record determination as to whether FITBONE is recommended. The decision to treat, observe, and to include in this observation study is at the discretion of the healthcare provider. This is an observational study and therefore, the participating healthcare provider will manage patients according to the usual clinical practice.

Surgery will be performed according to the standard surgical procedure described previously. Study of Investigational Product(s). Five to ten days after the lengthening nail placement, the lengthening mechanism is operated by transmitting energy necessary for the lengthening from the outside. This period is referred to as the distraction period. The rhythm of lengthening and strict protocol for an individual patient, indicating the daily lengths of lengthening to be applied, are decided by the healthcare provider taking into account all influencing factors. Therefore, the end of the distraction period, bone healing, implant removal, and 6 months post-implant removal may differ by individual. In the event the distraction period is extended by the healthcare provider, the new distraction period will determine the end of the distraction time point. All patients will be followed until the end of the scheduled study period regardless of any change in their treatment or other conditions.

Six visits are planned:

1. Surgery (baseline)
2. End of the distraction phase
3. End of bone healing
4. Implant removal
5. 6-month post-removal
6. 24-month post-surgery The satisfaction will be assessed at implant removal, 6 months post implant removal, and 24 months post-surgery.

The QoL will be assessed at baseline, at 6 months post implant removal, and 24 months post-surgery.

Pain will be assessed at all timepoints. Measurement of pain at the end of the distraction phase, the patient will be requested to report the pain experienced in the past week, at the moment, and during or immediately after the distraction period. At other time points, pain for only at the moment will be captured.

Range of motion (ROM) will be measured at the end of bone healing, and at the 24 months post-surgery.

Lengthening achieved will be measured at the end of bone healing. Any incidence of adverse events will be recorded at any point during the 24-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥12 years old, with congenital or acquired lower limb discrepancy greater than 30mm, undergoing femoral or tibia bone lengthening with FITBONE
* Patients with a regular indication for a surgical intervention with FITBONE according to manufacturer IFU
* The patient (or his/her legally acceptable representative) is capable of understanding the content of the Informed Consent Form (ICF)
* The informed consent form is correctly obtained

Exclusion Criteria:

* Patients with a medical condition that is contraindicated according to the FITBONE instruction for use.
* Patients with any conditions that, in the Investigator's opinion, may interfere with the study execution, including those likely to be lost to follow-up.
* Patients who have any conditions or medical condition that, in the investigator's opinion, may interfere with the study's execution or in which the patient should not participate for safety reasons.
* Patients requiring the application of or have already in-situ concomitant devices that cannot be safely removed (except for permitted concomitant devices).
* Patients participating in other clinical or have taken part in any clinical study in the last 3 months.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The aim of the study is to have a representative population of FITBONE patients in France, who are cimpliant with the inclusion criteria, during the 1 year enrollment period. Any centre in France that uses FITBONE in their routine clinical practice will be invited and have the opportunity to participate in this study. All centres must systematically and without exception offer every patient being implanted with FITBONE the opportunity to participate in the study, limiting selection bias and increasing the representativeness of this study to the French population.
Sampling Method: Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Describe Patients' Pain by Visual Analog Scale (VAS) | at 6 months after implant removal date and at 24 months follow-up
  Pain will be measured by the Pain by Visual Analog Scale (VAS), performed by the patient, through the Patient Global Evaluation Assessment and by the physician (Clinical Observer Global Assessment). The VAS for pain ranges from 0 to 10, with 0 representing no pain and 10 representing the worst imaginable pain.
Describe Patients' patient Quality of Life (QoL) using Short Form 36 Health Survey (SF-36) for adult patients and PedsQL (Pediatric Quality of Life Inventory) Generic Core Scale for children patients. | at 6 months after implant removal date and at 24 months follow-up
  The Quality of Life (QoL) will be measured by the Short Form 36 Health Survey (SF-36) or PedsQL (Pediatric Quality of Life Inventory) Generic Core Scale, depending on the patient's age at enrolment: SF-36 for adults and PedsQl for children. Short Form 36 Health Survey has two components: Physical Component Summary (PCS) Minimum 0, Maximum 100; Mental Component Summary (MCS) Minimum 0, Maximum 100. Higher scores on both the Physical and Mental Component Summary scales indicate a better outcome, reflecting better health-related quality of life. The PedsQL Generic Core Scales are scored on a scale of 0 to 100, with higher scores indicating better health-related quality of life and 0 represents the worst health-related quality of life.
Describe Patients' satisfaction | at 6 months after implant removal date and at 24 months follow-up
  A dedicated patients satisfaction questionnaire has been developed with key opinion leaders (KOLs) and expert groups on the limb leg discrepancy treatment. The satisfaction questionnaire is made of 5 questions, for each question the patient have to reply using the Patient Global Impression of change ranging from 1 to 7, with 1 representing Very much improved; to 7 being Very much worse.

SECONDARY OUTCOMES:
Monitor the clinical safety of Fitbone by collecting and characterizing the complications, expressed as adverse events and device deficiencies, associated with FITBONE | from surgery to 24 months follow-up
  The clinical safety of Fitbone will be measured Collecting and characterizing the complications (expressed as adverse events and device deficiencies) associated with FITBONE that will be assessed by the investigators.
Effectiveness of Fitbone by limb lengthening | at the end of bone healing, approximately 6 months
  The lengthening goal is considered 'achieved' when, at the end of bone healing, the limb length is within 5 mm of the lengthening objective defined by the investigator when using FITBONE.
Assess satisfaction evolution at implant removal , 6 months after Fitbone removal and at 24 months after surgery | from surgery to 24 months follow-up
  A dedicated patients satisfaction questionnaire has been developed with key opinion leaders (KOLs) and expert groups on the limb leg discrepancy treatment. The satisfaction questionnaire is made of 5 questions, for each question the patient have to reply using the Patient Global Impression of change ranging from 1 to 7, with 1 representing "Very much improved" to 7 being "Very much worse".
Describe evolution of QoL at 6 months after Fitbone removal and at 24 months after surgery, compared to baseline | from surgery to 24 months follow-up
  The Quality of Life (QoL) will be measured by the Short Form 36 Health Survey (SF-36) or PedsQL (Pediatric Quality of Life Inventory) Generic Core Scale, depending on the patient's age at enrolment: SF-36 for adults and PedsQl for children. Short Form 36 Health Survey has two components: Physical Component Summary (PCS) Minimum 0, Maximum 100; Mental Component Summary (MCS) Minimum 0, Maximum 100. Higher scores on both the Physical and Mental Component Summary scales indicate a better outcome, reflecting better health-related quality of life. The PedsQL Generic Core Scales are scored on a scale of 0 to 100, with higher scores indicating better health-related quality of life and 0 represents the worst health-related quality of life.
Describe pain at each visit using VAS | from surgery to 24 months follow-up
  Pain will be measured by the Pain by Visual Analog Scale (VAS), performed by the patient, through the Patient Global Evaluation Assessment and by the physician (Clinical Observer Global Assessment). The VAS for pain ranges from 0 to 10, with 0 representing no pain and 10 representing the worst imaginable pain.
Describe patients Range Of Motion (ROM in degrees) evolution at end of bone healing and at 24 months after surgery compared to baseline | from surgery to 24 months follow-up
  The knee range of motion will measured in degree Difference in the range of motion through the passive extension before surgery (baseline) to the end of bone healing, and at 24 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Franck Accadbled, Prof., Principal Investigator — Centre hospitalier universitaire (CHU) de Toulouse; Maxime Fabre-Aubrespy, MD, Principal Investigator — Hôpital Sainte-Marguerite AP-HM; Damien Fron, MD, Principal Investigator — CHU Lille; Jean-Christophe Ruzic, MD, Principal Investigator — CHU de La Réunion site Sud Saint-Pierre; Hassan Al Khoury Salem, MD, Principal Investigator — CHU de Saint-Étienne Hôpital Nord; Ludovic Paul Schneider, MD, Principal Investigator — CHU de Strasbourg
Locations (6):
- France (5):
  - CHU de Saint-Étienne Hôpital Nord, Saint-Etienne, Auvergne-Rhône-Alpes
  - CHU de Strasbourg, Strasbourg, Grand Est
  - CHU Lille - Hôpital Jeanne de Flandre, Lille, Hauts-de-France
  - Centre hospitalier universitaire (CHU) de Toulouse, Toulouse, Occitanie
  - Hôpital Sainte-Marguerite AP-HM, Marseille, Provence-Alpes-Côte d'Azur Region
- CHU de La Réunion site Sud Saint-Pierre, Saint-Pierre, La Réunion, Reunion